CLINICAL TRIAL: NCT00001323
Title: Neuropsychiatric Evaluation of Normal Subjects and Psychiatric and Neurologic Contrast Groups
Brief Title: Neuropsychiatric Evaluation of Healthy Volunteers and Adults With Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920262; 92-M-0262
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Brain Injury; Dementia; Healthy; Mental Disorder; Schizophrenia
Keywords: Cognition; Neuropsychology; Neuropsychological Tests; Neurological Exam; Psychiatric; Attention; Schizophrenic; Schizoaffective; Working Memory; Memory
MeSH Terms: conditions — Brain Injuries; Dementia; Mental Disorders; Schizophrenia

SUMMARY:
The purpose of this study is to evaluate the cognitive processes of participants with schizophrenia, participants with nervous system and mental disorders, and healthy volunteers.

Participants in this study will undergo cognitive tests of attention, memory, attention. Participants with attention deficit hyperactivity disorder (ADHD), traumatic brain injury (TBI), bipolar disorder, and Alzheimer's disease (AD) will be compared with participants with schizophrenia. A group of healthy adults and children will undergo cognitive tests to further delineate the degree of impairment in schizophrenia and neurological disorder participants.

DETAILED DESCRIPTION:
In this study, we propose to administer cognitive tests to schizophrenic patients and to neurologic patients who will serve as contrast groups for neuropsychological studies of patients with schizophrenia. These include studies of Alzheimers disease to dissociate size and organization of lexicon and ADHD to understand error patterns on CPT-type tests of attention and vigilance. However, the majority of studies will examine schizophrenia in relation to normal controls.

In addition, we propose to obtain test results from a local sample of normal subjects of varying ages and educational backgrounds to further delineate degree of impairment in these clinical groups. As well as assessing adults we wish to assess normal children. In particular, we wish to identify in children the size of their lexicon and their degree of semantic organization within their lexicon.

ELIGIBILITY:
INCLUSION CRITERIA

English-speaking adults between ages 21 to 65, in good health and free from significant substance abuse.

Children between ages 4 to 20 must not have a history of special education, using psychotropic medication in long-term counseling or with a history of seizures, head injury or CNS infections.

Normal controls will be recruited and screened for exclusionary morbidity by interview (e.g., no history of contact with mental health professionals, no history of diagnosable alcohol and/or substance abuse).

Normal controls will be recruited from building employees, local universities, from NIMH rosters, and the general public.

EXCLUSION CRITERIA

Excluded are adults with histories of dementing illness, movement disorder, affective disorders, developmental and/or acquired brain injury. Diagnoses will be made by review of medical records, interview, examination, and in the case of psychiatric diagnoses, a structured interview by SCID.

Advertisement will make clear that the subjects will be asked questions about family psychiatric history and their own history or psychiatric disorder, substance abuse, and neurological disease. Only if the subject answers these negatively will he or she participate in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 810
Dates: Start 1992-08; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldberg TE, Weinberger DR, Berman KF, Pliskin NH, Podd MH. Further evidence for dementia of the prefrontal type in schizophrenia? A controlled study of teaching the Wisconsin Card Sorting Test. Arch Gen Psychiatry. 1987 Nov;44(11):1008-14. doi: 10.1001/archpsyc.1987.01800230088014. PMID 3675128
- [Background] Seidman LJ. Schizophrenia and brain dysfunction: an integration of recent neurodiagnostic findings. Psychol Bull. 1983 Sep;94(2):195-238. No abstract available. PMID 6356196
- [Background] Weinberger DR, Berman KF, Zec RF. Physiologic dysfunction of dorsolateral prefrontal cortex in schizophrenia. I. Regional cerebral blood flow evidence. Arch Gen Psychiatry. 1986 Feb;43(2):114-24. doi: 10.1001/archpsyc.1986.01800020020004. PMID 3947207